CLINICAL TRIAL: NCT00154362
Title: A Multi-center, Randomized, Double-blind, Cross-over, Placebo-controlled Clinical Trial to Evaluate Efficacy and Safety of Oxcarbazepine p.o. (300-1200 mg/Day) as Adjuvant Therapy for Impulsivity and Aggressive Behavior in Conduct Disorders in Adolescents
Brief Title: The Efficacy and Safety of Oral Oxcarbazepine 300-1200 mg/Day as Adjuvant Therapy in the Treatment of Adolescents With Impulsivity and Aggressive Behavior in Conduct Disorder This Study is Not Being Conducted in the United States.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CTRI476BES04
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Conduct Disorder
Keywords: Oxcarbazepine, conduct disorder, adolescents
MeSH Terms: conditions — Conduct Disorder | interventions — Oxcarbazepine

INTERVENTIONS:
Drug: Oxcarbazepine

SUMMARY:
Conduct disorder is a group of psychiatric symptoms that can include clinical characteristics of impulsivity and aggressive behavior. This study will investigate the efficacy a safety of oxcarbazepine in the treatment of adolescents with conduct disorder.

ELIGIBILITY:
Inclusion Criteria:

* History of conduct disorder, oppositional defiant disorder, and disruptive behavior disorder not otherwise specified
* Score >8 on the Impulsivity Rating Scale

Exclusion Criteria:

* Other serious medical or psychiatric conditions excluding conduct disorder, oppositional defiant disorder, and disruptive behavior disorder not otherwise specified
* Treatment with antiepileptic medications

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2003-04; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Percentage reduction on Impulsivity Rating Scale (IRS)

SECONDARY OUTCOMES:
Percent reduction in the Modified Overt Aggression Scale (MOAS)

CONTACTS AND LOCATIONS:
Overall Officials: Celso Arango, MD, Principal Investigator — Hospital Gregorio Marañón,Madrid, Spain